CLINICAL TRIAL: NCT07093853
Title: Residual Ridge Changes in Mandibular Overdentures Retained by Four Locator Attachments Versus Four-Implant Bar Attachments: A 10-Year Retrospective Study
Brief Title: Mandibular Overdentures Retained by Four Locator Attachments Versus Four-Implant Bar Attachments
Status: Recruiting | Type: Observational
Sponsor: Menoufia University (Other)
Collaborators: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohammed El-Sawy, Dr, Menoufia University
Other Study IDs: ADMNF-00925
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Bone Loss
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I - Locator Attachments: Patients received four implants were placed in the lateral incisor and first premolar regions. Overdentures were retained using unsplinted Locator attachments, processed chairside via direct intraoral pick-up, with vent holes to allow resin escape. These prostheses were implant-retained and tissue-supported.
  Interventions: Other: Four Locator Attachments, Four Bar Attachment System
- Group II - Bar Attachments: Patient also received four implants in the same quadrilateral distribution. The implants were splinted with a custom-milled titanium bar, and overdentures were retained using clip attachments. These prostheses were designed to be fully implant-supported, minimizing soft tissue loading.
  Interventions: Other: Four Locator Attachments, Four Bar Attachment System

INTERVENTIONS:
Other: Four Locator Attachments, Four Bar Attachment System — This study retrospectively evaluated two types of implant-retained mandibular overdenture attachment systems placed in edentulous patients over a 10-year period. All patients received four dental implants placed in the interforaminal region (lateral incisor and first premolar areas).
  In the Locator group, each implant was restored with an individual Locator attachment, allowing for independent retention and easier hygiene access.
  In the Bar group, the four implants were splinted together with a rigid metal bar, and the overdenture was attached using clips that engaged the bar, offering splinted support and enhanced load distribution.
  Both interventions were designed to support mandibular overdentures and were compared in terms of their long-term effects on posterior mandibular ridge resorption, marginal bone loss around implants, and anterior maxillary ridge resorption.

SUMMARY:
This 10-year retrospective study investigates residual ridge changes in edentulous patients treated with mandibular overdentures (ODs) retained by either four Locator attachments or a four-implant bar system. Although two-implant ODs are well established, four-implant configurations may offer enhanced stability and function. Locator and bar attachments are commonly used, but their long-term effects on bone resorption patterns-especially posterior mandibular and anterior maxillary resorption-remain unclear. By standardizing implant positions, this study aims to directly compare the two systems to help guide clinicians in selecting the most effective attachment type for long-term success.

DETAILED DESCRIPTION:
Implant-supported mandibular overdentures (ODs) have become the preferred treatment for edentulous patients, particularly after the endorsement of this approach by the McGill and York consensus statements. Although the use of two implants is well established, emerging research supports the use of four implants to enhance denture stability, improve masticatory function, and better maintain the surrounding oral structures.

Among the available attachment systems, Locator and bar-retained attachments are the most frequently utilized, each offering specific benefits. Locator attachments are known for their simplicity, affordability, and ease of maintenance. In contrast, bar-retained systems provide more rigid splinting between implants and more even stress distribution. These systems differ biomechanically, especially regarding their impact on bone resorption in the posterior mandible, which plays a vital role in denture retention and function.

While some research has compared different attachment types, few studies have standardized implant number and position. Moreover, there is a lack of long-term comparative studies assessing four-implant mandibular ODs using both Locator and bar attachments. Critical outcomes such as posterior mandibular ridge resorption (PMandRR), marginal bone loss (MBL), and anterior maxillary ridge resorption (AMaxRR) must be examined to evaluate the long-term effectiveness and biomechanical performance of these attachment systems.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous mandible and maxilla for at least 12 months.
* Four interforaminal dental implants placed in the lateral incisor and first premolar regions.
* Opposing maxillary complete denture constructed using a muco-compressive impression technique, with maximum denture base extension and lingualized occlusion.
* Mandibular bone height between 15-25 mm at the symphysis region as measured on panoramic radiograph.
* Minimum 10-year follow-up with adequate radiographic documentation.

Exclusion Criteria:

* Systemic diseases affecting bone metabolism.
* Parafunctional habits (e.g., bruxism).
* Smokers of more than 10 cigarettes/day or those with alcohol abuse.
* Patients with implant failures, missing follow-up data, or implants placed outside the interforaminal region.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consisted of completely edentulous patients who received mandibular overdentures retained by four dental implants placed in the interforaminal region. Patients were selected retrospectively based on having been treated with either four Locator attachments or a four-implant bar attachment system and followed for a minimum period of 10 years. All participants had similar implant positioning (lateral incisor and first premolar areas) and were free from systemic conditions that could affect bone healing or implant success. Inclusion criteria required good oral hygiene compliance and regular follow-up records. Exclusion criteria included uncontrolled systemic diseases, history of head and neck radiation, and lack of long-term follow-up data.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss (MBL) | 10 years
  Crestal bone loss around dental implants

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed El-Sawy, PhD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Dentistry, Al Mansurah, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request from the corresponding author